CLINICAL TRIAL: NCT04103762
Title: Interest of Intravenous Cholangiography With Indocyanine Green, Compared to Contrast Cholangiography, in the Context of Laparoscopic Cholecystectomy for Grade 1 and 2 Acute Gallstone Cholecystitis: Prospective, Monocentric, Randomized Study
Brief Title: Interest of Intravenous Cholangiography With Indocyanine Green in the Context of Laparoscopic Cholecystectomy for Grade 1 and 2 Acute Gallstone Cholecystitis
Acronym: VIFCAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2017_843_0020
Record Dates: First submitted 2019-09-19; First posted 2019-09-25 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Lithiasis; Cholecystitis, Acute; Cholangiopathy
Keywords: acute lithiasis cholecystitis; intraoperative cholangiography; indocyanine green; cholecystectomy
MeSH Terms: conditions — Lithiasis; Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- indocyanine green (Experimental): During the surgery, intraoperative cholangiography using indocyanine green will be performed
  Interventions: Procedure: laparoscopic cholecystectomy; Diagnostic Test: systematic intraoperative cholangiography
- standard cpo (Active Comparator): During the surgery, intraoperative cholangiography using a contrast product "gold standard" will be performed
  Interventions: Procedure: laparoscopic cholecystectomy; Diagnostic Test: systematic intraoperative cholangiography

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy — laparoscopic cholecystectomy
Diagnostic Test: systematic intraoperative cholangiography — systematic intraoperative cholangiography in both groups (use of Indocyanine Green in ICG group and Iomeron in the CPO group)

SUMMARY:
Acute lithiasis cholecystitis (ALC) is the third most common cause of surgical emergency admission. The initial treatment of ALC associates a medical support and a cholecystectomy, preferentially performed laparoscopically in the first 5 days of evolution. During the surgery, intraoperative cholangiography (CPO) using a contrast product is the "gold standard" to identify the bile ducts. However CPO is performed in approximately 30% of laparoscopic cholecystectomy.

Laparoscopic cholecystectomy for ALC is associated with an increase in the rate of biliary ducts injuries compared with cholecystectomy for symptomatic vesicular lithiasis, evaluated at 0.8 % versus 0.1 %. Its higher rate is related to local inflammation that alters the biliary anatomy and complicates the identification of the bile ducts. Indocyanine green facilitates the visualization of extrahepatic biliary structures, which could reduce the risk of biliary wound and shorten the operating time.

ELIGIBILITY:
Inclusion Criteria:

* Adults patient (>18 years old)
* Patients requiring laparoscopic cholecystectomy for grade 1 or 2 acute gallstone cholecystitis according to Tokyo recommendations confirmed by radiological morphological examination
* Acute lithiasis cholecystitis (ALC) evolving for less than 5 days
* Patients affiliated to a social security scheme

Exclusion Criteria:

* Antecedent of biliary tract surgery
* Antecedent of cholecystectomy
* Contraindication to laparoscopy
* Contraindication to surgery
* Cholecystectomy by laparotomy out of hand
* Grade 3 cholecystitis according to Tokyo recommendations
* Acute alithiasis cholecystitis
* Cirrhosis
* Conversion for gangrenous ALC
* Patient with an allergy to indocyanine green
* Pregnant or lactating woman, childbearing age without effective contraception
* Minor patient
* Physical or psychological state that does not allow participation in the study, patient under guardianship or curatorship or patient deprived of liberty by a judicial or administrative decision (according with articles L 1121-6 and L 1121-8 of the French Public Health Code)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Change of surgical procedure after Indocyanine green injection | day 0 = the day of the surgery
  Change of surgical procedure after Indocyanine green injection compared to intraoperative cholangiography (CPO) using a contrast product as the "gold standard" to identify the bile ducts.
  Indocyanine green facilitates the visualization of extrahepatic biliary structures, which could reduce the risk of biliary wound and shorten the operating time.

SECONDARY OUTCOMES:
Comparison of CPO (intraoperative cholangiography) achievement rates with visualized rates of the main bile duct via indocyanine green | day 0 = the day of the surgery
  Comparison of CPO (intraoperative cholangiography) achievement rates with visualized rates of the main bile duct via indocyanine green
Comparison of biliary element recognition rate during laparoscopic cholecystectomy between CPO (intraoperative cholangiography) group and Indocyanine green injection (ICG) group before dissection | day 0 = the day of the surgery
  Comparison of biliary element recognition rate during laparoscopic cholecystectomy between CPO (intraoperative cholangiography) group and Indocyanine green injection (ICG) group before dissection
Comparison of biliary element recognition rate during laparoscopic cholecystectomy between CPO (intraoperative cholangiography) group and Indocyanine green injection (ICG) group after dissection | day 0 = the day of the surgery
  Comparison of biliary element recognition rate during laparoscopic cholecystectomy between CPO (intraoperative cholangiography) group and Indocyanine green injection (ICG) group after dissection

CONTACTS AND LOCATIONS:
Overall Officials: Osama ABOU ARAB, MD, Principal Investigator — CHU Amiens; Emilie Dumange Chapuis-Roux, MD, Principal Investigator — CHU Amiens; Ralucar Macovei, MD, Principal Investigator — CHU Amiens; Baptiste Brac, MD, Principal Investigator — CHU Amiens; Aurélien Gracient, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Defives H, Chive E, Diouf M, Ammar-Khodja N, Pellegrin A, Werey F, Yvart-Degardin J, Sabbagh C, Regimbeau JM. Value of intravenous cholangiography with indocyanine green during laparoscopic cholecystectomy for grade I or II acute lithiasic cholecystitis: Results of a prospective, open, randomized, monocentric study (VIFCAL trial). Curr Probl Surg. 2025 Aug;69:101788. doi: 10.1016/j.cpsurg.2025.101788. Epub 2025 May 2. No abstract available. PMID 40716885